CLINICAL TRIAL: NCT06671782
Title: Improving Patient Involvement in Care-A Pilot Study of a Comprehensive Pelvic Floor Muscle Exercise Program Before and After Radical Prostatectomy to Prevent Urinary Leakage
Brief Title: A Study of a Pelvic Floor Muscle Exercise Program Before and After Radical Prostatectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-212
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: Urinary incontinence; Pelvic Floor Muscle Exercise
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence | interventions — Biofeedback, Psychology; Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled pilot study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (usual care) (Active Comparator): Consented patients randomized to the control group will receive usual care at MSK. This will comprise standardized verbal (and sometimes also written) instructions about Kegel exercises from the nurse and/or urologist before the operation. All patients will complete the Prostate Quality of Life Survey at baseline and at 1.5, 3, and 6 months after radical prostatectomy (within ±2 weeks is considered acceptable to avoid protocol violations). This is part of the standard of care for patients undergoing prostatectomy.
  Interventions: Other: Kegel exercises; Other: Questionnaires
- intervention group (PFME program with biofeedback) (Experimental): Consented patients randomized to the intervention group will be referred to SPEAR Physical Therapy to undergo the study PFME training program. The team at SPEAR Physical Therapy regularly sees patients undergoing radical prostatectomy and is specially trained in PFME training for male patients. Patients in the intervention arm will undergo PFME training with a physical therapist 2 times before surgery (4-6 weeks [in person] and 3-4 weeks [in person], before surgery) (within ±1 week is considered acceptable to avoid protocol violations). Patients in the intervention group will also undergo 2 PFME training sessions after surgery (3 weeks and 1.5 months after surgery).
  Interventions: Other: Pelvic Floor Muscle Exercise Program with biofeedback; Other: Questionnaires; Other: Interviews

INTERVENTIONS:
Other: Kegel exercises — Kegel exercises without any formal training
  Arms: control group (usual care)
Other: Pelvic Floor Muscle Exercise Program with biofeedback — Patients in the intervention arm will undergo PFME training with a physical therapist 2 times before surgery (4-6 weeks [in person] and 3-4 weeks [in person], before surgery) (within ±1 week is considered acceptable to avoid protocol violations). Patients in the intervention group will also undergo 2 PFME training sessions after surgery (3 weeks and 1.5 months after surgery).
  Arms: intervention group (PFME program with biofeedback)
Other: Questionnaires — All patients will complete the Prostate Quality of Life Survey at baseline and at 1.5, 3, and 6 months after radical prostatectomy (within ±2 weeks is considered acceptable to avoid protocol violations). This is part of the standard of care for patients undergoing prostatectomy.
Other: Interviews — A qualitative interview with each of the 15 patients in the intervention group to obtain information about the patient's experience. The interview will last for 30-60 min and will be conducted at 3-6 months after prostatectomy, when the patient has completed all 4 physical therapy sessions. It will cover topics related to patient involvement, satisfaction, and activation.
  Arms: intervention group (PFME program with biofeedback)

SUMMARY:
The researchers are doing this study to find out if a PFME program to reduce urinary incontinence after radical prostatectomy is feasible for people with prostate cancer. The researchers will track how many participants join the study, follow the program, and stay in the study. They will also evaluate how people feel about their experience and satisfaction with participating in this program through interviews. They will also measure participants' quality of life by filling out questionnaires, and we will study whether the program shows promise in reducing urinary incontinence.

Radical prostatectomy sometimes causes incontinence after the surgery. The researchers think that by teaching PFME and strengthening and improving control of the pelvic floor muscles, PFME training before and after radical prostatectomy may help reduce incontinence and/or reduce how long incontinence lasts.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years with prostate cancer scheduled for radical prostatectomy at MSK

Exclusion Criteria:

* Previous radiotherapy for prostate cancer
* Urinary incontinence at baseline before radical prostatectomy
* Inability to participate in study activities (exercise program, imaging, and questionnaires) because of:

  * Comorbidity(-ies) and/or
  * Geographic location and/or
  * Communication barrier(s)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 32 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Assessing rate of accrual | up to six months after surgery
  Assess the feasibility of a comprehensive, physical therapist-instructed pre- and postoperative PFME program by determining rates of accrual

CONTACTS AND LOCATIONS:
Overall Officials: James Eastham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm